CLINICAL TRIAL: NCT03877575
Title: Lyon Uveitis Study
Acronym: LYS
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2019_003
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No specific intervention. Collection of clinical data

SUMMARY:
Uveitis or inflammation of the uveal tract results from a heterogeneous collection of disorders of varying etiologies and pathogenic mechanisms. Uveitis is relatively frequent in industrial countries with an estimation of 115 cases for 100 000 persons and is associated with a blindness risk of 10%. Causes of uveitis can be related to different etiologies (infectious, inflammatory or general inflammatory diseases). Therapeutic care is based on ophthalmologic and systemic diagnosis and treatment strategy depends on the severity of inflammation.

The main objective of the Lyon uveitis study is to analyze the uveitis ophthalmologic etiology and diagnostic and therapeutic care of the patients. This study is proposed to all patients diagnosed for uveitis and referred to the Department of Internal Medicine of the Croix Rousse hospital, Lyon, france for etiologic diagnosis or treatment.

Analysis of i) patients' characteristics, ii) the relevance of complementary exams to determine the uveitis etiology, iii) treatment used.

This study will allow a better characterization of the disease on diagnosis practices and therapeutic care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uveitis
* First consultation in the Department of Internal Medicine at the Croix-Rousse hospital, Lyon, France

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is proposed to all patients diagnosed for uveitis and referred to the Department of Internal Medicine of the Croix-Rousse hospital, Lyon, France for the first visit corresponding to etiologic diagnosis or treatment.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical evolution (persistence or resolution) evaluated by gradation of SEN | At one year after diagnosis
  Persistence of disease is characterized by persistence of intraocular inflammation evaluated by gradation of SEN. (reference: A Standardization Grading System for Scleritis . Ophthalmology 2011 Apr;118(4):768-71). SEN score ranges from 0 to 5 (resolution = score 0 and persistence = score >0)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No